CLINICAL TRIAL: NCT00617825
Title: Cryotherapy for Chronic Venous Disorders
Brief Title: Feasibility Study of Cryotherapy for Chronic Venous Disorders
Acronym: Cryo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Teresa J. Kelechi, PhD, RN, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17504; 1R21NR010604-01 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2007-09

CONDITIONS: Venous Insufficiency
Keywords: chronic venous disorders; cryotherapy; skin microcirculation; skin temperature
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: cyrotherapy as a cool gel wrap — A cool gel wrap made of a hydrogel with silicon will be applied to the lower leg of skin affected by venous disorders for 30 minutes each day for 30 days during the study
  Other Names: Elastogel Therapy Wrap

SUMMARY:
Severe skin damage caused by chronic venous disorders (CVDs) results in relentless pain and poor quality of life for millions of adults in the U.S. each year. DVDs are under-recognized and under-treated disorders shat harm the veins of the legs and at worst, cause skin inflammation and venous leg ulcers. A new way to ease the pain and inflammation is proposed in this study of cryotherapy (cool gel wraps) applied to damaged skin of the lower legs of CVD-affected individuals. The study hypothesis predicts that this novel cryotherapy model and method will significantly improve the health and quality of life for those with CVDs and that the intervention will become a standard of care for CVDs. In addition, the method will, over time, reduce health care costs associated with treating poor CVD outcomes.

DETAILED DESCRIPTION:
Chronic venous disorders (CVDs) often cause long-term disability for those who experience the worst manifestations of CVDs: disabling pain and non-healing leg ulcers. Such disabilities have significant socioeconomic implications in terms of lost work days and wages, decreased productivity,and ultimately increased health care costs that deteriorate the well-being and quality of life for those who have CVD-induced illnesses. Because no reliable preventive mechanisms exists for CVDs, this study proposes a preventive, self-management cryotherapy intervention that targets inflamed skin of populations with CVDs at highest risk of developing chronic leg ulcers. The proposed cryotherapy intervention will utilize a randomized controlled clinical trial to develop a method to reduce clinical symptoms by improving existing therapy - it is not a treatment for CVDs itself. In the proposed pilot feasibility study, subjects will be randomized to two groups; the cryotherapy intervention group (n=30) who will receive a four-week, cryotherapy gel wrap applied daily to the affected skin of the lower legs in addition to the standard of care (usual care). The control group (n=30) will receive the usual care of compression wraps or stockings applied to the lower legs and daily leg elevation. With this method, improvement of skin microcirculation, reduced leg pain, and improvement in quality of life will be observed. The following aims will test the hypothesis:

Aim 1: Evaluate the feasibility of the novel intervention including treatment fidelity, subject training, safety, and side effects associated with equipment and recruitment efforts and further refine the intervention protocol, including questionnaires used in our previous studies.

Aim 2: Estimate variability of outcome measurements and effect sizes needed to calculate sample size for a subsequent larger, adequately powered, randomized clinical trial of the efficacy of the novel cryotherapy intervention.

Aim 3: Investigate the presence of a preliminary "signal" of clinical efficacy of the experimental treatment by evaluating trends toward statistical significance for the hypothesis that the experimental group will experience greater reduction in skin temperature and blood flow, greater improvement in pain, and greater improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 years and older
* CEAP classification: stage C4 (changes in skin and subcutaneous tissue secondary to CVDs)4a (pigmentation or eczema) 4b (lipodermatosclerosis or atrophie blanche) C5 (healed venous ulcers)
* Ankle brachial index (ABI) 0.9 - 1.3mm Hg 0 absence of peripheral arterial disease
* Intact skin sensation measured with 10 gram monofilament
* Intact thermal sensation measured with thermal sensory tester at lower leg skin and foot surfaces
* Agreement to wear compression garments such as wraps or stockings during waking hours
* Phone, e-mail, or mail accessible
* Working freezer

Exclusion Criteria:

* ABI < 0.8 mm Hg or > 1.3 mm Hg -presence of lower extremity arterial disease (reduces skin temperature)
* Active systemic or localized infections such as cellulitis (raises skin temperature)
* Autoimmune disorders that reduce blood flow such as Raynaud's phenomenon
* Body temperature > 37.6 degrees C (febrile state raises skin temperature)
* CEAP classification c6: active venous ulcer (cooling ulcerated skin might impair healing)
* Known peroneal nerve injury
* Impaired skin sensation
* Unable to detect light touch measured with a 10 gram monofilament at lower leg skin surfaces
* Unable to detect not/cold sensation measured with thermal sensory tester at lower leg skin surfaces
* Not wearing compression or not agreeing to wear compression wraps or stockings
* Phone, e-mail, or mail inaccessible
* No working freezer

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
improvement of skin microcirculation | 30 days

SECONDARY OUTCOMES:
leg pain | 30 days
quality of life | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kelechi, PhD, RN, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States